CLINICAL TRIAL: NCT01851109
Title: Prevention of Ovarian Cancer in Women Participating in Mammography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Swedish Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R18DP001142-01 (NIH)
Record Dates: First submitted 2013-05-03; First posted 2013-05-10 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Epithelial Ovarian Cancer
Keywords: ovarian cancer; prevention; prophylactic surgery; risk; biomarkers; screening; symptoms
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Ovarian Neoplasms | interventions — Genetic Counseling

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention)
- Genetic counseling (Experimental): After randomization the participant is offered a referral to a genetic counselor.
  Interventions: Behavioral: genetic counseling

INTERVENTIONS:
Behavioral: genetic counseling — The genetic counseling sessions are conducted by a licensed genetic counselor, certified by the American Board of Genetic Counseling and the American Board of Medical Genetics. This clinical counseling session may include, but is not limited to the following:
  1. A review of medical and family history information to determine which genetic test (BRCA, HNPCC, p53, etc.), if any, is appropriate;
  2. Discuss how the results - positive or negative - affect cancer risk
  3. Discuss how cancer risk might be managed (surveillance, prophylactic surgery, oral contraceptives, etc.);
  4. Discuss how the test is conducted and what the results might be (positive, negative, uncertain);
  5. Discuss the disadvantages of genetic testing (cost, insurance coverage, worry about insurance discrimination, uncertain results, etc.) and the psychological and emotional issues surrounding testing, etc.
  Arms: Genetic counseling

SUMMARY:
The primary purpose of this study is to evaluate the effect of systematic identification and genetic counseling referral on rates of bilateral salpingo-oophorectomy (surgery to remove both fallopian tubes and ovaries) in women having mammograms at Swedish Medical Center in Seattle, WA.

ELIGIBILITY:
Inclusion Criteria:

* Prior mammogram at Swedish Medical Center
* Willing and able to provide informed consent, primary physician information, and complete study questionnaires
* Must meet at least ONE of the following criteria:
* personal history of breast cancer diagnosed before age 50
* personal history of bilateral breast cancer at any age
* 1 or more first degree relatives with breast cancer diagnosed before age 50
* 3 or more first or second degree relatives with breast cancer at any age
* 2 second degree relatives with breast cancer diagnosed before age 50
* A male relative with breast cancer at any age
* Ashkenazi Jewish with any family history of breast or ovarian cancer
* 1 first or second degree relative with ovarian cancer AND 1 first or second degree relative with breast cancer at any age
* 2 first degree relatives with ovarian cancer or 2 second degree relatives with ovarian cancer or 1 first and 1 second degree relative with ovarian cancer.
* A first degree relative with both breast and ovarian cancer (2 primaries in the same person)
* Personal history of positive genetic test result for any of the following genes: BRCA1, BRCA2, HNPCC, or P53
* Family history of a positive genetic test result for any of the following genes: BRCA1, BRCA2 or HNPCC

Exclusion Criteria:

* Previous diagnosis of ovarian cancer
* Prior bilateral-salpingo oophorectomy
* Had a negative genetic test result for a known family genetic mutation

Min Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2008-07; Primary Completion 2013-05 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Compare rates of risk-reducing salpingo-oophorectomy in each of the study arms | 24 months post-enrollment

SECONDARY OUTCOMES:
Cancer related distress | change from baseline at 12 and 24 months post-enrollment
Health-related quality of life | change from baseline at 12 and 24 months post-enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Urban, ScD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States